CLINICAL TRIAL: NCT04105608
Title: A Mediterranean-pattern Meal Increases GLP-1 and Oxyntomodulin More Than an Energy-matched High Fiber Plant-Based Meal in Type 2 Diabetes Patients: A Randomized Clinical Trial Assessment Through the Visual Analogue Scale.
Brief Title: GLP-1 and Oxyntomodulin Release in Relation to Diet in Type 2 Diabetes Patients.
Acronym: VAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Antonio Di Mauro (Other)
Responsible Party: Sponsor-Investigator, Antonio Di Mauro, Registered Dietitian Nutritionist, Campus Bio-Medico University
Organization: Campus Bio-Medico University (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 08/2017
Record Dates: First submitted 2019-09-23; First posted 2019-09-26 (Actual); Last update posted 2019-09-26 (Actual); Status verified 2019-09

CONDITIONS: Type-2 Diabetes
Keywords: Diabetes; GLP-1; Oxyntomodulin; Diet; Visual Analogue Scale
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HFV meal (Experimental): A vegetarian meal high in dietary carbohydrate and fiber
  Interventions: Dietary Supplement: High-fiber vegetarian meal
- MED meal (Active Comparator): A Mediterranean-like meal
  Interventions: Dietary Supplement: Mediterranean-like meal

INTERVENTIONS:
Dietary Supplement: High-fiber vegetarian meal — The intervention consisted in the administration of a high fiber vegetarian meal prepared by our research group staff.
  Arms: HFV meal
Dietary Supplement: Mediterranean-like meal — The intervention consisted in the administration of a Mediterranean-like meal prepared by our research group staff.
  Other Names: Control meal
  Arms: MED meal

SUMMARY:
The aim of this trial was to assess glycemic control and incretin release in subjects affected by type-2 diabetes, a condition in which GLP-1 release is impaired. It is known that nutrition affects a variety of factors in overall quality of life in diabetes and we hypothesized incretin secretion may improve in acute. As little is known regarding oxyntomodulin secretion in relation to diet, we explored this gut-derived hormone behavior as well.

Hence, the administration of two meals was carried out; these were equal in terms of calories but different for macronutrients composition. Appetite rating was assessed as well through a 100-mm horizontal Visual Analogue Scale, either at fasting and for 4 hours once the meal was completed.

DETAILED DESCRIPTION:
Type-2 diabetes (T2D) is a multifactorial metabolic burden whose metabolic features include alterations in GLP-1 secretion and ultimately hunger/satiety circuit derangement. Manipulating the composition of the diet in order to promote GLP-1 secretion may represent a promising lifestyle strategy for obesity and T2D management.

The objective of this study was to assess the post-prandial profile of appetite- regulating hormones and assessing the post-prandial appetite ratings using a Visual Analogue Scale (VAS), as well as measuring the fasting and postprandial glucose/insulin responses in overweight and/or obese, well controlled patients with T2D.

Twelve T2D patients (M:F = 7:5) aged 63.1±8.5 years were enrolled in a randomized, controlled, crossover trial. Subjects consumed on two different days, at one-week interval, an experimental High Fiber Vegetarian meal (HFV) rich in dietary carbohydrate and fiber in comparison with a standard, Mediterranean-like meal (MED). The two meals were isocaloric. Appetite ratings, glucose/insulin and gastrointestinal hormone responses were assessed either at fasting and every 30' until 210' for GLP-1 and Oxyntomodulin and 240' for glucose and insulin after the ingestion of the meal.

ELIGIBILITY:
Inclusion Criteria:

* Type-2 diabetes history of at least 2 years, age above 18 years, body mass index (BMI) between 25 and 35 kg/m2, and drug naïve and/or with metformin treatment.

Exclusion Criteria:

* clinically significant neurological, endocrinological, or other systemic diseases, as well as those with acute illness and chronic inflammatory or infective disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — 1:1
Enrollment: 12 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2017-12-01 (Actual); Study Completion 2018-02-28 (Actual)

PRIMARY OUTCOMES:
Changes in serum GLP-1 concentration | 0' (fasting), +30', +60', +90', +120', +150', +180, +210', +240' (minutes)
  Changes in serum GLP-1 levels following the ingestion of the two meals

SECONDARY OUTCOMES:
Changes in plasma oxyntomodulin concentration | 0' (fasting), +30', +60', +90', +120', +150', +180, +210', +240' (minutes)
  Plasma oxyntomodulin assessment in relation to HFV and MED meal.
Serum glucose and insulin levels | 0' (fasting), +30', +60', +90', +120', +150', +180, +210', +240' (minutes)
  Serum blood glucose and insulin levels
Hunger-satiety scores (millimeters) | 0' (fasting), +30', +60', +90', +120', +150', +180, +210', +240' (minutes)
  We assessed VAS scores in relation to meals through the quantification of self-reported hunger, satiety, and desire to eat. Participants were asked to mark a validated 10-mm horizontal scale (Visual analogue scale) at multiple time points [0' (fasting), +30', +60', +90', +120', +150', +180, +210', +240' (minutes)]. These ratings were subsequently quantified and assessed for potential correlation with any of the hormones assessed (i.e., GLP-1, oxyntomodulin, glucose, and insulin). Each scale had a left end equal to zero mm (i.e., "not at all") and a right end equal to 100 mm (i.e., "absolutely" or "definitely yes"), with no subscales. Each participant was instructed on how to fill the questionnaire properly and every assessment occurred with no disturbance and/or any other patient.

CONTACTS AND LOCATIONS:
Locations (1):
- Campus Bio-Medico University of Rome, Rome, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Di Mauro A, Tuccinardi D, Watanabe M, Del Toro R, Monte L, Giorgino R, Rampa L, Rossini G, Kyanvash S, Soare A, Rosati M, Piccoli A, Napoli N, Fioriti E, Pozzilli P, Khazrai YM, Manfrini S. The Mediterranean diet increases glucagon-like peptide 1 and oxyntomodulin compared with a vegetarian diet in patients with type 2 diabetes: A randomized controlled cross-over trial. Diabetes Metab Res Rev. 2021 Sep;37(6):e3406. doi: 10.1002/dmrr.3406. Epub 2020 Sep 24. PMID 32926502